CLINICAL TRIAL: NCT04051424
Title: A Pilot Study in Healthy Volunteers of McKay Airway - An Improved Oral Airway for Awake Fibre-optic Intubation
Brief Title: New Airway for Awake Intubation (McKay Airway)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, William McKay, M.D., University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BIO 17 - 202
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Design: The proposed experiment is a randomized clinical crossover (repeated measures) trial of three oral bite-block devices with device order randomized and blinded prior to recruitment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ConMed bite block (Active Comparator): Standard bite block (Conmed Bite Block; Conmed Corp., Utica NY, USA)
  Interventions: Device: McKay airway; Device: Williams Airway
- Williams Airway (Active Comparator): Williams Airway Intubator (Williams Airway Intubator Ltd, Calgary, Canada)
  Interventions: Device: ConMed bite block; Device: McKay airway
- McKay airway (Experimental): A new device that enables maintenance of jaw thrust. (US patent application 16/098,530)
  Interventions: Device: ConMed bite block; Device: Williams Airway

INTERVENTIONS:
Device: ConMed bite block — Investigator will fit ConMed bite block in patient's mouth and bronchoscopist will try to visualize the vocal cords.
  Arms: McKay airway; Williams Airway
Device: McKay airway — Investigator will fit McKay airway in patient's mouth and bronchoscopist will try to visualize the vocal cords.
  Arms: ConMed bite block; Williams Airway
Device: Williams Airway — Investigator will fit Williams Airway in patient's mouth and bronchoscopist will try to visualize the vocal cords.
  Arms: ConMed bite block; McKay airway

SUMMARY:
When endotracheal intubation is known or predicted to be difficult, patients are intubated awake using a flexible bronchoscope (awake fibre-optic intubation: AFI) so that they can protect their airway with normal upper airway muscle activity until the endotracheal tube (ETT) is safely in place. New bite blocks have been invented for bag mask ventilation but are not suitable for AFI.1 A newly invented airway device, the McKay airway, may provide a better solution for AFI by enabling jaw thrust, a condition where the upper airway is opened more as the jaw is protruded forward. It may also be more comfortable for awake users. A study is proposed to assess the functionality of the device for this purpose.

To protect the bronchoscope, a bite block is used during AFI to protect the very delicate glass fibres from damage from inadvertent biting by the patient. Currently used bite blocks protect the scope, but do not position the jaw optimally for scoping. The proposed device is an attempt to improve upon current bite blocks by both protecting the bronchoscope and positioning the jaw optimally.

Hypothesis: Residents in training in the Division of Respirology have limited experience in fibre-optic bronchoscopy and perform it under the direct supervision of an expert. Null hypothesis: the time to visualization of vocal cords with a fibre-optic bronchoscope by residents learning in the Division of Respirology will be no different with the McKay airway than with the conventional bite block or Williams Airway.

DETAILED DESCRIPTION:
INTRODUCTION When endotracheal intubation is known or predicted to be difficult, patients are intubated awake using a flexible bronchoscope so that they can protect their airway with normal upper airway muscle activity until the endotracheal tube (ETT) is safely in place. A newly invented airway device, the McKay airway, (Appendix 2) may provide a better solution to placing an ETT into the windpipe of an awake patient, (awake fibre-optic intubation: AFI) A study is proposed to assess the functionality of the device for this purpose.

To protect the bronchoscope, a bite block is used during AFI to protect the very delicate glass fibres from damage from inadvertent biting by the patient. Currently used bite blocks (Appendix 2, figure 5) protect the scope, but do not position the jaw or bronchoscope optimally for scoping. This is not a problem for experienced bronchoscopists such as respirologists, but can be for those, like anesthesiologists, who do bronchoscopy infrequently. For these, the proposed device may be an improvement upon current bite blocks.

Hypothesis: Residents in training in the Division of Respirology have limited experience in fibre-optic bronchoscopy and perform it under the direct supervision of an expert. Null hypothesis: the time to visualization of vocal cords with a fibre-optic bronchoscope by residents learning in the Division of Respirology will be no different with the McKay airway than with the conventional bite block.

Experimental design: The proposed experiment is an unblinded repeated measures interventional clinical trial with concealed randomization of which device is used first and which second. Randomization will be by a computer-generated random number table (1s and 2s where 1 is conventional bite block is used first and 2 means McKay airway first) transcribed to paper cards in numbered opaque envelopes to be opened just prior to bronchoscopy.

Primary outcome: Time from beginning insertion of bronchoscope into the bite block to visualization of vocal cords.

Secondary outcomes: Scores will be recorded on rating scales for: ease of insertion, ease of obtaining proper position of teeth in the device by patients, assessment of gag reflex. Comments about overall impression will be recorded.

Participants: Participants are of two kinds, patients and residents. Patients will be consenting patients booked for bronchoscopy by pulmonologists at Royal University Hospital. Excepted patients will be those who do not wish to participate and those with any health conditions that the attending pulmonologist feels puts them at any added risk by participating.

Consent: With University of Saskatchewan Research Ethics Board approval, the investigators will recruit patients and obtain signed informed consent at the time of booking bronchoscopy or on arrival for bronchoscopy.

Data and privacy concerns: As well as the primary and secondary outcomes, data collection on paper data sheets will include basic demographics. These are: age, gender, height, weight, and diagnosis as well as airway characteristics (see Appendix 1, Data Sheet). Because this may identify patients and breach their privacy, the data sheets will be identified only by number. The de-identified data collection sheets will be labeled with a unique numerical identifier (e.g., 1, 2, 3, etc). The data collection sheet will be linked to the patient Personal Health Number by way of a physically separate Master Data list (e.g., 1, 2, 3, etc.). (See attached - Master Data List) The de-identified data from the data collection sheet (See Attached - Data Collection Sheet) will be transcribed by Dr. McKay to data base on a password protected computer kept in a locked office in the Department of Anesthesiology at all times. Identifiable patient information will not be transcribed electronically. Upon completion of the study, Dr McKay will store electronic data files and paper forms in a locked filing cabinet in the Department of Anesthesiology (accessible only by key code), as per the University of Saskatchewan Research Integrity Policy (http://www.usask.ca/university_secretary/policies/research/8_25.php). The Master Data List (paper only) will be stored in a physically separate location from the data collection forms. The hard copies of the data collection forms, master list, and completed consent forms will be destroyed through the confidential paper disposal services of the SHR, while the electronic data will be permanently deleted after 5 years as per the above University of Saskatchewan Research Integrity Policy. We anticipate this data to be the basis for a publication in a peer-reviewed scientific journal and at a national scientific meeting.

Patient safety: The experiment will be overseen by the attending specialist respirologist who will intervene immediately as needed and proceed as clinically indicated if any issue of patient safety arises at any time. This is normal practice. We expect that risk to participating patients is minimal. We anticipate the following incidence: 1) common (1-10%) side effects: none. 2) uncommon (0.1 to 1%) side effects: mild abrasion of the mouth (which can occur with the currently available awake intubation bite blocks and airways as often). 3) rare (0.01-0.1%) side effects: zero. 4) Very rare (<0.01%) side effects: sensitivity to the plastic with irritation of the oral mucosa (which can occur with the currently available awake intubation plastic bite blocks and airways as often). The McKay airway is made of medical grade plastic. 5) Severe side effects: zero (prolonged hospital admission, admission to intensive care, loss of limb or vital organ, or death). We believe that risk of participation is not different from risk of bronchoscopy, and is safe in expert hands.

Measurements. With a stopwatch, the investigator will measure the time from beginning to place the bronchoscope in the mouth following topicalization to visualization of vocal cords or epiglottis. Following bronchoscopy, the Respirologist will rate the modalities with rating scales (see attached Data Sheet).

Number of participants: There is no similar study from which to calculate sample size. We will initially assuming that one modality is 0.2 times faster with standard deviation 0.2, paired t-test sample size is calculated at n = 10, then recalculate based on the primary outcome findings.

Statistical analysis. Demographic and rating data will be tabulated as observational; time measurements compared by paired t-test or Mann-Whitney U test as mean ± standard deviation and [95% Confidence Intervals] or median and [interquartile range] as appropriate following a Kolmogorov-Smirnov test of normality.

ELIGIBILITY:
Inclusion Criteria:

* Participants are of two kinds, first, anesthesiologists and anesthesia residents who will perform partial bronchoscopy, and
* secondly, healthy volunteers. Healthy volunteers will be recruited from hospital staff, residents and students at Royal University Hospital.

Exclusion Criteria:

* Excepted anesthesiologists and residents will be those who do not wish to participate in the study.
* Excepted volunteers will be those who do not wish to participate in the study and those with a lidocaine allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Ease of use. | 5 minutes
  Ordinal scale comparison with standard bite block for ease of obtaining a bronchoscopic view of vocal cords or epiglottis (scale of 1 to 5 - see data sheets below).
Time to visualize cords. | 5 minutes
  Time in seconds from starting bronchoscope insertion to cord visualization.

SECONDARY OUTCOMES:
Usefulness. | 5 minutes
  Ordinal scale comparison with standard bite block (scale of 1 to 5 - see data sheets below) for: ease of insertion, ease of obtaining proper position of teeth in the device by patients, assessment of gag reflex, and likelihood of employing the method in practice. Comments about overall impression will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: William P McKay, MD, Principal Investigator — Professor Emeritus
Locations (1):
- Saskatoon Health Region, 410 22nd Street East, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data (all) will be available from Dr McKay - email request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: June 2017 - indefinitely
Access Criteria: Interested applicant